CLINICAL TRIAL: NCT05217446
Title: A PHASE 2, RANDOMIZED, OPEN-LABEL STUDY OF ENCORAFENIB AND CETUXIMAB PLUS PEMBROLIZUMAB VERSUS PEMBROLIZUMAB ALONE IN PARTICIPANTS WITH PREVIOUSLY UNTREATED BRAF V600E-MUTANT, MSI H/DMMR METASTATIC COLORECTAL CANCER
Brief Title: A Study of Encorafenib Plus Cetuximab Taken Together With Pembrolizumab Compared to Pembrolizumab Alone in People With Previously Untreated Metastatic Colorectal Cancer
Acronym: SEAMARK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Merck KGaA, Darmstadt, Germany (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4221022; SEAMARK (Other: Alias Study Number); 2024-512119-34-00 (Registry Identifier: CTIS (EU)); KEYNOTE-D31 (Other: Merck); MK-3475-D31 (Other: Merck)
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Keynote-D31; BRAF V600E mutation positive; Colon cancer; Rectal cancer; Metastatic colon cancer; Colon cancer BRAF; Rectal cancer BRAF; MSI-H colorectal cancer; MSI-H colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — encorafenib; Cetuximab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter study of encorafenib and cetuximab plus pembrolizumab (Triplet Arm [Arm A]) versus pembrolizumab alone (Control Arm [Arm B]) as first-line treatment in participants with BRAF inhibitor (BRAF) V600E-mutant and microsatellite instability-high/ deficient mismatch repair (MSI-H/dMMR) mCRC. Randomization will be stratified by ECOG (0 vs 1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: encorafenib, cetuximab and pembrolizumab (Experimental): Participants receive encorafenib orally + cetuximab IV + pembrolizumab IV.
  Interventions: Drug: Encorafenib; Biological: Cetuximab; Biological: Pembrolizumab
- Arm B: pembrolizumab (Active Comparator): Participants receive pembrolizumab IV.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Drug: Encorafenib — capsule
  Other Names: PF-07263896 LGX818 ONO-7702 W0090
  Arms: Arm A: encorafenib, cetuximab and pembrolizumab
Biological: Cetuximab — IV
  Other Names: Erbitux
  Arms: Arm A: encorafenib, cetuximab and pembrolizumab
Biological: Pembrolizumab — IV
  Other Names: Keytruda®, MK-3475

SUMMARY:
The purpose of this study is to learn about the effects of three study medicines (encorafenib, cetuximab, and pembrolizumab) given together for the treatment of colorectal cancer that:

* is metastatic (spread to other parts of the body);
* has the condition of genetic hypermutability (tendency to mutation) or impaired DNA mismatch repair (MMR)
* has a certain type of abnormal gene called "BRAF" and;
* has not received prior treatment.

All participants in this study will receive pembrolizumab at the study clinic as an intravenous (IV) infusion (given directly into a vein) at the study clinic.

In addition, half of the participants will take encorafenib by mouth at home every day and cetuximab by IV infusion at the study clinic.

The study team will monitor how each participant is doing with the study treatment during regular visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

* Locally confirmed microsatellite instability-high/ deficient mismatch repair (MSI-H/dMMR) stage IV colorectal carcinoma
* Locally confirmed BRAF V600E mutation in tumor tissue or blood
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have not received prior systemic regimens for metastatic disease.
* Measurable disease per RECIST 1.1
* Adequate organ function

Exclusion Criteria:

* Colorectal adenocarcinoma that is RAS mutant or for which RAS mutation status is unknown
* Known active central nervous system metastases and/or carcinomatous meningitis; leptomeningeal disease
* Immunodeficiency or active autoimmune disease requiring systemic treatment in the past 2 years
* Presence of acute or chronic pancreatitis
* Clinically significant cardiovascular diseases (eg, thromboembolic or cerebrovascular accident events ≤ 12 wks prior)
* Received a live or live-attenuated vaccine within 30 days of planned start of study medication
* Previous treatment with any selective BRAF inhibitor (eg, encorafenib, dabrafenib, vemurafenib, XL281/BMS-908662) or any epidermal growth factor receptor (EGFR) inhibitor (eg, cetuximab, panitumumab).
* Previous treatment with an immune checkpoint inhibitor (eg, anti-programmed cell death [PD-1], anti-PD-L1 or anti-PD-L2 agent); or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Duration of study, approximately 45 months
  PFS per investigator, defined as the time from randomization until PD based on investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurs first:

SECONDARY OUTCOMES:
Incidence of adverse events | Duration of study, approximately 45 months
  Incidence and severity of AEs graded according to the NCI CTCAE v4.03: encorafenib and cetuximab + pembrolizumab (Arm A) vs pembrolizumab (Arm B)
Overall Survival (OS) | Duration of study, approximately 45 months
  OS is defined as the time from the date of randomization to the date of death due to any cause: encorafenib and cetuximab + pembrolizumab (Arm A) vs pembrolizumab (Arm B)
Objective Response (OR) | Duration of study, approximately 45 months
  OR is defined as a CR or PR per RECIST version 1.1 recorded from the date of randomization until date of first documentation of PD, death, or start of new anti-cancer therapy: encorafenib and cetuximab + pembrolizumab (Arm A) vs pembrolizumab (Arm B)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (6):
  - Mayo Clinic Building - Phoenix, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Mount Sinai Cancer Center, Miami Beach, Florida
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (3):
  - Imelda General Hospital, Bonheiden, Antwerpen
  - Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-capitale, Région de
- Canada (3):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences - Odette Cancer Centre, Toronto, Ontario
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice Bulovka, Prague, Praha 8
- Denmark (4):
  - Rigshospitalet, Copenhagen, Capital Region
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
  - Vejle Sygehus, Vejle, Region Syddanmark
- France (5):
  - Hôpital Européen Georges Pompidou, Paris, Paris
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - CHU Estaing, Clermont-Ferrand
  - Institut Regional du Cancer de Montpellier - ICM Val d'Aurelle, Montpellier
  - Hôpital Saint Antoine, Paris
- Germany (2):
  - Muenchen Klinik Neuperlach, Klinik fuer Haematologie und Onkologie, Munich, Bavaria
  - Facharztzentrum Eppendorf, Hamburg
- Italy (12):
  - Policlinico Universitario Monserrato, Monserrato, Cagliari
  - Azienda Ospedaliera Universitaria dell'Università "Luigi Vanvitelli" Piazza Luigi Miraglia, 2 Napoli, Napoli, Campania
  - Ospedale di Guastalla, Guastalla, Emilia-Romagna
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Azienda USL Toscana Nord Ovest_Ospedale Civile di Livorno, Livorno, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Arcispedale Santa Maria Nuova, Reggio Emilia
- Maastricht UMC+, Maastricht, Limburg, Netherlands
- Oslo Universitetssykehus Ullevål, Oslo, Norway
- Poland (2):
  - Przychodnia Lekarska KOMED, Konin, Greater Poland Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów
- Narodny onkologicky ustav, Bratislava, Slovakia
- Spain (9):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen CITY
  - Heartlands Hospital, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Elez E, Kopetz S, Tabernero J, Bekaii-Saab T, Taieb J, Yoshino T, Manji G, Fernandez K, Abbattista A, Zhang X, Morris VK. SEAMARK: phase II study of first-line encorafenib and cetuximab plus pembrolizumab for MSI-H/dMMR BRAFV600E-mutant mCRC. Future Oncol. 2024 Apr;20(11):653-663. doi: 10.2217/fon-2022-1249. Epub 2023 Oct 10. PMID 37815847
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221022